CLINICAL TRIAL: NCT00094575
Title: CSP #498 - Open Versus Endovascular Repair (OVER) Trial for Abdominal Aortic Aneurysms
Brief Title: Standard Open Surgery Versus Endovascular Repair of Abdominal Aortic Aneurysm (AAA)
Acronym: OVER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 498
Record Dates: First submitted 2004-10-20; First posted 2004-10-21 (Estimated); Results first posted 2013-12-31 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Aortic Aneurysm
Keywords: Abdominal; Aortic Aneurysm; cost of AAA repair; Endovascular Repair; Grafts; Long-term survival; secondary outcomes
MeSH Terms: conditions — Aortic Aneurysm | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): Standard Open Repair of Abdominal Aortic Aneurysm
  Interventions: Procedure: Standard Open Repair
- Arm 2 (Active Comparator): Endovascular Repair of Abdominal Aortic Aneurysm
  Interventions: Procedure: Endovascular Repair

INTERVENTIONS:
Procedure: Endovascular Repair — Endovascular Repair
  Arms: Arm 2
Procedure: Standard Open Repair — Standard Open Repair
  Arms: Arm 1

SUMMARY:
A multi-center, randomized clinical trial that will compare endovascular repair with standard open surgery in the repair of abdominal aortic aneurysms (AAA). Long and short-term results as well as the cost and quality of life associated with these two strategies for AAA repair will be compared.

DETAILED DESCRIPTION:
Primary Hypothesis: All-cause mortality will differ by 25% between Endovascular repair (EVR) and Open repair. Secondary Hypotheses: Procedure failure, short term (12-month) major morbidity, number of hospital days, health-related quality of life and other procedure-related abnormalities will differ between the two AAA repair strategies. Primary Outcomes: All-cause mortality. Interventions: Patients will be randomized to one of these repair strategies for the elective treatment of AAA: (a) Open repair or (b) Endovascular repair (using FDA-approved devices). Study Abstract: Aortic aneurysm is the tenth leading cause of death in older men; AAA accounts for the majority of these deaths (about 10,000 deaths per year in the United States). Since one in 22 Veterans over the age of 50 have AAA and one in 200 have AAA with diameter greater or equal to 5.0 cm (making them candidates for elective repair), AAA is a major disease in the VA population. Questions about the relative safety and effectiveness of FDA approved EVR devices have been raised and remain unanswered. To answer these questions, this multi-center, randomized clinical trial comparing EVR with standard open surgery is proposed. Patients for whom elective repair of AAA is indicated and who are suitable candidates for both open repair and EVR will be eligible for the study. The anticipated duration of the study is 9 years with a proposed sample size of 900 patients. The first planning meeting took place on March 9-10, 2000 and the second planning meeting took place on November 6-7, 2000. The OVER protocol was submitted and reviewed by CSEC on May 10, 2001 and approved. The kickoff was June 12, 2002. The first DSMB meeting took place January 6, 2003. First annual meeting was held September 30, 2003; second DSMB meeting took place September 29, 2003. Third DSMB meeting held on April 19, 2004; second annual meeting was held on June 29, 2004. Fourth DSMB meeting was held on December 6, 2004; third annual meeting was held on March 15, 2005. The fifth DSMB meeting was held on July 19, 2005 and the fourth annual meeting was held March 21, 2006. The sixth DSMB meeting was held September 12, 2005. The seventh DSMB meeting was held on March 6, 2006. The eighth DSMB meeting was held on November 6, 2006. At its November 6, 2006 meeting, the DSMB discussed and approved unblinding of the study chair to prepare the short-term follow-up paper as specified in the study protocol. Initially the protocol called for this analysis to include one-year follow-up data. After discussions with the Trial Leadership, the DSMB approved use of two year follow-up data (reflected in DSMB minutes finalized February 20, 2007). This recommendation was subsequently approved by CSP in March 2007. The short-term outcomes manuscript was published in JAMA on October 14, 2009. The ninth DSMB meeting was held on May 14, 2007 and the fifth annual meeting was held on June 6, 2007. The tenth DSMB meeting was held on April 7, 2008. The eleventh DMC (name change only from DSMB to DMC) was held on June 22, 2009. The twelfth DMC meeting was held on May 24, 2010. A Site Investigator meeting was held in Boston, MA on June 9, 2010. The thirteenth DMC meeting was held on June 3, 2011 and a study close-out meeting was held on June 15, 2011 in Chicago, IL. The study's patient follow-up phase ended October 15, 2011.

ELIGIBILITY:
Inclusion Criteria:

* AAA with a maximum external diameter in any plane greater than or equal to 5 cm.
* An iliac aneurysm (associated with an AAA) with a maximum external diameter in any plane greater than or equal to 3 cm.
* AAA greater than or equal to 4.5 cm and the AAA has increased by greater than or equal to 0.7 cm in diameter in 6 months.
* An AAA greater than or equal to 4.5 cm and the AAA has increased by greater than or equal to 1 cm in diameter in 12 months.
* An AAA greater than or equal to 4.5 cm and the AAA is saccular (i.e., a portion of the circumference of the aorta at the level of the aneurysm is considered normal based on CT scan or MRI).
* An AAA greater than or equal to 4.5 cm and the AAA is associated with distal embolism.

  * as measured from two imaging studies (ultrasound CT scan or MRI) within the appropriate interval, the later one within 6 months of randomization.

Exclusion Criteria:

* Patient has had a previous AAA repair procedure
* Evidence of AAA rupture by imaging test
* AAA is not elective (i.e., urgent or emergent operation, usually due to suspected rupture)
* Likelihood of poor compliance to the protocol
* Patient refused randomization
* Physician refused randomization

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 881 (Actual)
Dates: Start 2002-10; Primary Completion 2011-10 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank A. Lederle, MD, Study Chair — Minneapolis Veterans Affairs Medical Center
Locations (42):
- United States (42):
  - VA Medical Center, Birmingham, Birmingham, Alabama
  - Southern Arizona VA Health Care System, Tucson, Tucson, Arizona
  - Central Arkansas VHS Eugene J. Towbin Healthcare Ctr, Little Rock, No. Little Rock, Arkansas
  - VA Medical Center, Loma Linda, Loma Linda, California
  - VA Medical Center, Long Beach, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, San Diego, California
  - VA Medical Center, San Francisco, San Francisco, California
  - VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California
  - VA Eastern Colorado Health Care System, Denver, Denver, Colorado
  - VA Connecticut Health Care System (West Haven), West Haven, Connecticut
  - VA Medical Center, DC, Washington D.C., District of Columbia
  - North Florida/South Georgia Veterans Health System, Gainesville, Florida
  - James A. Haley Veterans Hospital, Tampa, Tampa, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia
  - Jesse Brown VAMC (WestSide Division), Chicago, Illinois
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - Richard Roudebush VA Medical Center, Indianapolis, Indianapolis, Indiana
  - VA Medical Center, Iowa City, Iowa City, Iowa
  - VA Medical Center, Lexington, Lexington, Kentucky
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland
  - VA Boston Healthcare System, Brockton Campus, Brockton, Massachusetts
  - John D. Dingell VA Medical Center, Detroit, Detroit, Michigan
  - Minneapolis VA Health Care System, Minneapolis, Minnesota
  - VA Medical Center, Omaha, Omaha, Nebraska
  - VA New Jersey Health Care System, East Orange, East Orange, New Jersey
  - New Mexico VA Health Care System, Albuquerque, Albuquerque, New Mexico
  - VA Western New York Healthcare System at Buffalo, Buffalo, New York
  - New York Harbor HCS, New York, New York
  - VA Medical Center, Durham, Durham, North Carolina
  - VA Medical Center, Cincinnati, Cincinnati, Ohio
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - VA Medical Center, Portland, Portland, Oregon
  - VA Medical Center, Philadelphia, Philadelphia, Pennsylvania
  - VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania
  - VA Medical Center, Memphis, Memphis, Tennessee
  - VA North Texas Health Care System, Dallas, Dallas, Texas
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, Salt Lake City, Utah
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington
  - Wlliam S. Middleton Memorial Veterans Hospital, Madison, Madison, Wisconsin
  - Zablocki VA Medical Center, Milwaukee, Milwaukee, Wisconsin

REFERENCES:
- [Result] Lederle FA. Vascular disease: is AAA screening worth the cost? Nat Rev Cardiol. 2009 Oct;6(10):616-8. doi: 10.1038/nrcardio.2009.161. No abstract available. PMID 19773791
- [Result] Lederle FA, Freischlag JA, Kyriakides TC, Padberg FT Jr, Matsumura JS, Kohler TR, Lin PH, Jean-Claude JM, Cikrit DF, Swanson KM, Peduzzi PN; Open Versus Endovascular Repair (OVER) Veterans Affairs Cooperative Study Group. Outcomes following endovascular vs open repair of abdominal aortic aneurysm: a randomized trial. JAMA. 2009 Oct 14;302(14):1535-42. doi: 10.1001/jama.2009.1426. PMID 19826022
- [Result] Dalainas I. Comparing endovascular and open repair of abdominal aortic aneurysm. JAMA. 2010 Feb 10;303(6):513; author reply 514. doi: 10.1001/jama.2010.86. No abstract available. PMID 20145222
- [Result] Lederle FA. The rise and fall of abdominal aortic aneurysm. Circulation. 2011 Sep 6;124(10):1097-9. doi: 10.1161/CIRCULATIONAHA.111.052365. No abstract available. PMID 21900095
- [Result] Lederle FA. The strange relationship between diabetes and abdominal aortic aneurysm. Eur J Vasc Endovasc Surg. 2012 Mar;43(3):254-6. doi: 10.1016/j.ejvs.2011.12.026. Epub 2012 Jan 9. PMID 22237512
- [Result] Stroupe KT, Lederle FA, Matsumura JS, Kyriakides TC, Jonk YC, Ge L, Freischlag JA; Open Versus Endovascular Repair (OVER) Veterans Affairs Cooperative Study Group. Cost-effectiveness of open versus endovascular repair of abdominal aortic aneurysm in the OVER trial. J Vasc Surg. 2012 Oct;56(4):901-9.e2. doi: 10.1016/j.jvs.2012.01.086. Epub 2012 May 27. PMID 22640466
- [Result] Lederle FA, Freischlag JA, Kyriakides TC, Matsumura JS, Padberg FT Jr, Kohler TR, Kougias P, Jean-Claude JM, Cikrit DF, Swanson KM; OVER Veterans Affairs Cooperative Study Group. Long-term comparison of endovascular and open repair of abdominal aortic aneurysm. N Engl J Med. 2012 Nov 22;367(21):1988-97. doi: 10.1056/NEJMoa1207481. PMID 23171095
- [Result] Lederle FA, Stroupe KT; Open Versus Endovascular Repair (OVER) Veterans Affairs Cooperative Study Group. Cost-effectiveness at two years in the VA Open Versus Endovascular Repair Trial. Eur J Vasc Endovasc Surg. 2012 Dec;44(6):543-8. doi: 10.1016/j.ejvs.2012.10.002. Epub 2012 Oct 30. PMID 23116986
- [Result] Lederle FA. Abdominal aortic aneurysm: still no pill. Ann Intern Med. 2013 Dec 17;159(12):852-3. doi: 10.7326/0003-4819-159-12-201312170-00012. No abstract available. PMID 24490269
- [Result] Lal BK, Zhou W, Li Z, Kyriakides T, Matsumura J, Lederle FA, Freischlag J; OVER Veterans Affairs Cooperative Study Group. Predictors and outcomes of endoleaks in the Veterans Affairs Open Versus Endovascular Repair (OVER) Trial of Abdominal Aortic Aneurysms. J Vasc Surg. 2015 Dec;62(6):1394-404. doi: 10.1016/j.jvs.2015.02.003. PMID 26598115
- [Derived] Lederle FA, Kyriakides TC, Stroupe KT, Freischlag JA, Padberg FT Jr, Matsumura JS, Huo Z, Johnson GR; OVER Veterans Affairs Cooperative Study Group. Open versus Endovascular Repair of Abdominal Aortic Aneurysm. N Engl J Med. 2019 May 30;380(22):2126-2135. doi: 10.1056/NEJMoa1715955. PMID 31141634
- [Derived] Powell JT, Sweeting MJ, Ulug P, Blankensteijn JD, Lederle FA, Becquemin JP, Greenhalgh RM; EVAR-1, DREAM, OVER and ACE Trialists. Meta-analysis of individual-patient data from EVAR-1, DREAM, OVER and ACE trials comparing outcomes of endovascular or open repair for abdominal aortic aneurysm over 5 years. Br J Surg. 2017 Feb;104(3):166-178. doi: 10.1002/bjs.10430. PMID 28160528
- [Derived] Lederle FA, Stroupe KT, Kyriakides TC, Ge L, Freischlag JA; Open vs Endovascular Repair (OVER) Veterans Affairs Cooperative Study Group. Long-term Cost-effectiveness in the Veterans Affairs Open vs Endovascular Repair Study of Aortic Abdominal Aneurysm: A Randomized Clinical Trial. JAMA Surg. 2016 Dec 1;151(12):1139-1144. doi: 10.1001/jamasurg.2016.2783. PMID 27627802
- [Derived] Myers SA, Applequist BC, Huisinga JM, Pipinos II, Johanning JM. Gait kinematics and kinetics are affected more by peripheral arterial disease than by age. J Rehabil Res Dev. 2016;53(2):229-38. doi: 10.1682/JRRD.2015.02.0027. PMID 27149635
- [Derived] Matsumura JS, Stroupe KT, Lederle FA, Kyriakides TC, Ge L, Freischlag JA; Open Versus Endovascular Repair (OVER) Veterans Affairs Cooperative Study Group. Costs of repair of abdominal aortic aneurysm with different devices in a multicenter randomized trial. J Vasc Surg. 2015 Jan;61(1):59-65. doi: 10.1016/j.jvs.2014.08.003. Epub 2014 Sep 16. PMID 25238728

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Repair: Standard Open Repair
Period: Overall Study
Arm/Group | Endovascular Repair | Open Repair
Started | 444 | 437
Completed | 298 | 291
Not Completed | 146 | 146
Not completed — Death | 146 | 146

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endovascular Repair | Open Repair | Total
Number analyzed (Participants) | 444 | 437 | 881
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (7.8) | 70.5 (7.8) | 70.1 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 441 | 435 | 876
Weight in kilograms [Mean (Standard Deviation); unit: Kilogram] | 89.9 (16.8) | 89.7 (17.8) | 89.8 (17.3)
Body Mass Index [BMI] [Mean (Standard Deviation); unit: Kg/m^2] | 28.6 (5.2) | 28.7 (5.6) | 28.6 (5.4)
Smoking Status [Number; unit: Participants]
  Ever Smoked | 428 | 413 | 841
  Never Smoked | 16 | 24 | 40
Currently Smoking [Number; unit: Participants]
  Yes | 170 | 193 | 363
  No | 274 | 244 | 518
Surgical Risk [RAND Score] [Number; unit: Participants]
  Low | 240 | 228 | 468
  Intermediate | 169 | 175 | 344
  High | 31 | 29 | 60
  Not Assessed | 4 | 5 | 9
Maximum Aneurysm Diameter [Mean (Standard Deviation); unit: Centimeter] | 5.7 (.8) | 5.7 (1.0) | 5.7 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality
Description: Participants vital status was assessed from randomization to end of study follow-up [10/15/2011] or death [whichever occurred first].
Time Frame: Participants were followed for the duration of the study, up to 9 years
Measure: Number; unit: participants
Arm/Group | Endovascular Repair | Open Repair
Number analyzed (Participants) | 444 | 437
participants | 146 | 146
Statistical Analysis 1: Comparison: Endovascular Repair vs Open Repair; The primary outcome was long-term, all-cause mortality. The sample size would provide 80% power to detect a 25% relative reduction in mortality at a two-sided alpha level of 0.05. The primary comparison was the main effects of Endovascular repair vs Open repair of AAA; Test type: Superiority or Other; p = 0.81, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.77 to 1.22] — The HR was estimated by comparing Endovascular repair arm vs the Open repair arm

2. Secondary Outcome: Secondary Therapeutic Procedures
Description: This outcome includes any procedure that resulted directly or indirectly from the initial procedure and that required a separate trip to the procedure suite (with each trip to the procedure suite counting as one secondary procedure), including any unplanned surgical procedures within 30 days after the initial procedure and any additional aortoiliac procedures at any time.
Time Frame: Participants were followed for the duration of the study, up to 9 years
Measure: Number; unit: participants
Arm/Group | Endovascular Repair | Open Repair
Number analyzed (Participants) | 444 | 437
participants | 98 | 78
Statistical Analysis 1: Comparison: Endovascular Repair vs Open Repair; Test type: Superiority or Other; p = 0.12, Chi-squared

3. Secondary Outcome: SF-36 Mental Component Score (MCS)
Description: Change (over time) since baseline in Mental Component Score of SF-36. The MCS Score ranges from 0-100 with higher scores indicating better health. Longitudinal mixed-effects model, adjusted for baseline values, was used to compare the two study arms. Treatment effect and change in quality-of-life measures over time were assessed in repeated measures models (with unstructured covariance) with the assigned repair method and baseline measurements used as covariates.
  Least-squares mean changes from baseline were calculated at each time point; the reported overall least squares mean is calculated over all time points.
Time Frame: Outcome was assessed at 6 months and then yearly, up to 9 years
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Endovascular Repair | Standard Open Repair
Number analyzed (Participants) | 444 | 437
units on a scale | -0.77 [-1.42 to -0.12] | -0.66 [-1.32 to 0.002]
Statistical Analysis 1: Comparison: Endovascular Repair vs Standard Open Repair; Test type: Superiority or Other; p = 0.81, Mixed Models Analysis

4. Secondary Outcome: SF-36 Physical Component Score (PCS)
Description: Change (over time) since baseline in Physical Component Score of SF-36. The PCS Score ranges from 0-100 with higher scores indicating better health Longitudinal mixed-effects model, adjusted for baseline values, was used to compare the two study arms. Treatment effect and change in quality-of-life measures over time were assessed in repeated measures models (with unstructured covariance) with the assigned repair method and baseline measurements used as covariates.
  Least-squares mean changes from baseline were calculated at each time point; the reported overall least squares mean is calculated over all time points.
Time Frame: Outcome was assessed at 6 months and yearly thereafter, up to 9 years
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Endovascular Repair | Standard Open Repair
Number analyzed (Participants) | 444 | 437
units on a scale | -3.18 [-3.91 to -2.45] | -3.05 [-3.79 to -2.31]
Statistical Analysis 1: Comparison: Endovascular Repair vs Standard Open Repair; Test type: Superiority or Other; p = 0.80, Mixed Models Analysis

5. Secondary Outcome: SF-36 Physical Component Deaths Included Score (PCTD)
Description: Change (over time) since baseline in Physical Component Deaths included Score of SF-36.
  The PCTD Score ranges from 0-100 with higher scores indicating better health. Longitudinal mixed-effects model, adjusted for baseline values, was used to compare the two study arms. Treatment effect and change in quality-of-life measures over time were assessed in repeated measures models (with unstructured covariance) with the assigned repair method and baseline measurements used as covariates.
  Least-squares mean changes from baseline were calculated at each time point; the reported overall least squares mean is calculated over all time points.
Time Frame: Outcome was assessed at 6 months and yearly thereafter, up to 9 years
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Endovascular Repair | Standard Open Repair
Number analyzed (Participants) | 444 | 437
units on a scale | -7.30 [-8.94 to -5.67] | -6.98 [-8.64 to -5.32]
Statistical Analysis 1: Comparison: Endovascular Repair vs Standard Open Repair; Test type: Superiority or Other; p = 0.78, Mixed Models Analysis

6. Secondary Outcome: European Quality of Life-5 Dimension (EQ-5D) Index Score
Description: Change (over time) since baseline in EQ-5D. The EQ-5D Index Score ('thermometer scale') ranges from 0 (worst health status) to 100 (best health status). Since this outcome captures change since baseline, values could be below 0.
  Longitudinal mixed-effects model, adjusted for baseline values, was used to compare the two study arms. Treatment effect and change in quality-of-life measures over time were assessed in repeated measures models (with unstructured covariance) with the assigned repair method and baseline measurements used as covariates.
  Least-squares mean changes from baseline were calculated at each time point; the reported overall least squares mean is calculated over all time points.
Time Frame: Outcome was assessed at 6 months and yearly thereafter, up to 9 years
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Endovascular Repair | Standard Open Repair
Number analyzed (Participants) | 444 | 437
units on a scale | -3.67 [-4.91 to -2.43] | -3.17 [-4.43 to -1.91]
Statistical Analysis 1: Comparison: Endovascular Repair vs Standard Open Repair; Note: Since this is measuring change over time since baseline, values could be below 0; Test type: Superiority or Other; p = 0.58, Mixed Models Analysis

7. Secondary Outcome: European Quality of Life-5 Dimension (EQ-5D) Visual Analog Scale
Description: Change (over time) since baseline in EQ-5D Visual Analog Scale. The EQ-5D Visual Analog Scale ranges from 0 (death) to 1 (perfect health). Longitudinal mixed-effects model, adjusted for baseline values, was used to compare the two study arms. Treatment effect and change in quality-of-life measures over time were assessed in repeated measures models (with unstructured covariance) with the assigned repair method and baseline measurements used as covariates.
  Least-squares mean changes from baseline were calculated at each time point; the reported overall least squares mean is calculated over all time points.
Time Frame: Outcome was assessed at 6 months and yearly thereafter, up to 9 years
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Endovascular Repair | Standard Open Repair
Number analyzed (Participants) | 444 | 437
units on a scale | -0.04 [-0.05 to -0.03] | -0.03 [-0.05 to -0.02]
Statistical Analysis 1: Comparison: Endovascular Repair vs Standard Open Repair; Test type: Superiority or Other; p = 0.37, Mixed Models Analysis

8. Secondary Outcome: International Index of Erectile Function (IIEF-5)
Description: Change (over time) since baseline in IIEF-5. The IIEF-5 Score ranges from 5-25 with higher scores indicating better erectile function.
  Longitudinal mixed-effects model, adjusted for baseline values, was used to compare the two study arms. Treatment effect and change in quality-of-life measures over time were assessed in repeated measures models (with unstructured covariance) with the assigned repair method and baseline measurements used as covariates.
  Least-squares mean changes from baseline were calculated at each time point; the reported overall least squares mean is calculated over all time points.
Time Frame: Outcome was assessed at 6 months and yearly thereafter, up to 9 years
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Endovascular Repair | Standard Open Repair
Number analyzed (Participants) | 444 | 437
units on a scale | -3.54 [-4.18 to -2.89] | -3.73 [-4.38 to -3.08]
Statistical Analysis 1: Comparison: Endovascular Repair vs Standard Open Repair; Test type: Superiority or Other; p = 0.68, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Endovascular Repair | Open Repair
Serious Adverse Events (participants affected / at risk) | 336/444 | 329/437
Other Adverse Events (participants affected / at risk) | 127/444 | 177/437
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular Repair (N=444) | Open Repair (N=437)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 8 (8)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 5 (5) | 9 (10)
Angina pectoris (Cardiac disorders) | 2 (2) | 3 (3)
Angina unstable (Cardiac disorders) | 2 (2) | 2 (2)
Arrhythmia (Cardiac disorders) | 0 (0) | 3 (4)
Arteriosclerosis coronary artery (Cardiac disorders) | 4 (4) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 16 (17) | 15 (19)
Atrial flutter (Cardiac disorders) | 4 (4) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 3 (3)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) | 5 (6)
Cardiac arrest (Cardiac disorders) | 4 (4) | 11 (11)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3) | 4 (4)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 23 (31) | 28 (44)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Chordae tendinae rupture (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 11 (14) | 9 (10)
Coronary artery occlusion (Cardiac disorders) | 6 (6) | 5 (5)
Coronary artery stenosis (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial infarction (Cardiac disorders) | 16 (18) | 23 (26)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial rupture (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular hypokinesia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 7 (13)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Cushing's syndrome (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Corneal degeneration (Eye disorders) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 5 (5)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 9 (9)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 3 (3)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 2 (2) | 2 (3)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4) | 6 (7)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 3 (3) | 4 (4)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 3 (5)
Inguinal hernia (Gastrointestinal disorders) | 2 (3) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 5 (6)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 5 (5)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric occlusion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 3 (3)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Post-tussive vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2)
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 (2) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 7 (8)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Adverse drug reaction (General disorders) | 3 (4) | 3 (3)
Asthenia (General disorders) | 2 (2) | 4 (4)
Cardiac death (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 17 (20) | 8 (11)
Death (General disorders) | 24 (24) | 14 (14)
Device dislocation (General disorders) | 4 (5) | 0 (0)
Device malfunction (General disorders) | 1 (1) | 2 (2)
Device occlusion (General disorders) | 2 (2) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1)
Hernia obstructive (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Medical device complication (General disorders) | 0 (0) | 3 (3)
Multi-organ failure (General disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 4 (4) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 2 (2)
Sudden cardiac death (General disorders) | 2 (2) | 0 (0)
Ulcer haemorrhage (General disorders) | 0 (0) | 1 (1)
Unevaluable event (General disorders) | 2 (2) | 3 (3)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 4 (4)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 6 (7)
Cholelithiasis (Hepatobiliary disorders) | 5 (5) | 4 (4)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 2 (2) | 0 (0)
Babesiosis (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 5 (7) | 5 (5)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 (0) | 1 (1)
Campylobacter intestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Cardiac valve vegetation (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 9 (9) | 9 (14)
Cellulitis orbital (Infections and infestations) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 4 (4) | 6 (6)
Device related infection (Infections and infestations) | 1 (1) | 2 (2)
Diverticulitis (Infections and infestations) | 5 (6) | 5 (6)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter sepsis (Infections and infestations) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 0 (0) | 1 (1)
Fungal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Graft infection (Infections and infestations) | 5 (6) | 1 (1)
Groin infection (Infections and infestations) | 10 (10) | 1 (1)
HIV infection (Infections and infestations) | 0 (0) | 2 (2)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Injection site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 2 (2)
Lobar pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection pseudomonal (Infections and infestations) | 2 (3) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (2)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 48 (61) | 37 (55)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 2 (2) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 3 (3) | 5 (6)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 3 (5)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (2) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 17 (19) | 18 (20)
Urosepsis (Infections and infestations) | 3 (3) | 2 (2)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Viral labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 4 (5)
Accidental exposure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Aortic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Confusion postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 27 (32) | 31 (38)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Graft complication (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Graft dysfunction (Injury, poisoning and procedural complications) | 21 (25) | 0 (0)
Graft thrombosis (Injury, poisoning and procedural complications) | 5 (7) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (3) | 9 (9)
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 6 (6) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Splenic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Urinary bladder rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 6 (7) | 1 (1)
Vascular injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vena cava injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 0 (0) | 1 (1)
Anticoagulation drug level below therapeutic (Investigations) | 0 (0) | 1 (1)
Arteriogram normal (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0)
Blood culture positive (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Bronchoscopy (Investigations) | 0 (0) | 1 (1)
Cardiac enzymes increased (Investigations) | 1 (1) | 0 (0)
Cardiac enzymes normal (Investigations) | 0 (0) | 1 (1)
Cardiac stress test abnormal (Investigations) | 1 (1) | 0 (0)
Colonoscopy (Investigations) | 1 (1) | 0 (0)
Computerised tomogram thorax abnormal (Investigations) | 1 (1) | 0 (0)
Diagnostic procedure (Investigations) | 0 (0) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1)
Heart rate irregular (Investigations) | 1 (1) | 0 (0)
Vitamin B12 decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 8 (9) | 8 (8)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
Adrenal gland cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Angiosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (3)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Laryngeal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 7 (8)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 5 (6)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (4)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Malignant mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Non-small cell lung cancer stage IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (6)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 3 (4)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 2 (2)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery disease (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 2 (2)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 18 (22) | 11 (12)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Complex partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 3 (5) | 3 (3)
Dementia (Nervous system disorders) | 1 (1) | 3 (3)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (2)
Lacunar infarction (Nervous system disorders) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 3 (3)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Spinal cord ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 10 (10) | 6 (7)
Syringomyelia (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 3 (4)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium tremens (Psychiatric disorders) | 0 (0) | 3 (3)
Impaired self-care (Psychiatric disorders) | 0 (0) | 1 (1)
Intentional drug misuse (Psychiatric disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 2 (2)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Schizoaffective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 3 (3)
Suicide attempt (Psychiatric disorders) | 0 (0) | 2 (2)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrogenic diabetes insipidus (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 4 (4) | 2 (2)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery occlusion (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 4 (4)
Renal failure acute (Renal and urinary disorders) | 10 (10) | 10 (10)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal ischaemia (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric dilatation (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Pelvic haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Priapism (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 23 (34) | 38 (62)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (6)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 12 (13)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Dry gangrene (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Homicide (Social circumstances) | 0 (0) | 1 (1)
Physical disability (Social circumstances) | 0 (0) | 1 (1)
Treatment noncompliance (Social circumstances) | 2 (2) | 2 (2)
Abdominal hernia repair (Surgical and medical procedures) | 0 (0) | 5 (5)
Alcohol detoxification (Surgical and medical procedures) | 0 (0) | 2 (2)
Anticoagulant therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Blood product transfusion (Surgical and medical procedures) | 0 (0) | 1 (1)
Carotid artery stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Carotid endarterectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 3 (3)
Colostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 2 (2) | 2 (3)
Coronary artery bypass (Surgical and medical procedures) | 2 (2) | 4 (4)
Diabetes mellitus management (Surgical and medical procedures) | 1 (1) | 0 (0)
Endotracheal intubation (Surgical and medical procedures) | 0 (0) | 2 (2)
Enteral nutrition (Surgical and medical procedures) | 0 (0) | 1 (1)
Extubation (Surgical and medical procedures) | 0 (0) | 1 (1)
Fluid replacement (Surgical and medical procedures) | 1 (1) | 1 (1)
Gastrostomy tube insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Haematoma evacuation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Ileostomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Incisional drainage (Surgical and medical procedures) | 1 (1) | 1 (1)
Leg amputation (Surgical and medical procedures) | 1 (1) | 1 (1)
Lung lobectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Rehabilitation therapy (Surgical and medical procedures) | 0 (0) | 2 (2)
Removal of foreign body (Surgical and medical procedures) | 0 (0) | 1 (1)
Self-medication (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Strangulated hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Tracheostomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Transurethral bladder resection (Surgical and medical procedures) | 1 (1) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 2 (2) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Ureteral stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Vascular stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Wound drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 2 (3) | 2 (2)
Aortic aneurysm rupture (Vascular disorders) | 4 (4) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 2 (2)
Arterial rupture (Vascular disorders) | 0 (0) | 1 (1)
Arterial stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 4 (4) | 7 (7)
Bloody discharge (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 5 (6) | 7 (8)
Femoral artery occlusion (Vascular disorders) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 3 (4)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 3 (3)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 2 (2) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Vascular disorders) | 0 (0) | 2 (2)
Ischaemia (Vascular disorders) | 3 (3) | 4 (5)
Ischaemic limb pain (Vascular disorders) | 0 (0) | 1 (1)
Lymphocele (Vascular disorders) | 1 (1) | 1 (1)
Microangiopathy (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 3 (3) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 3 (5)
Peripheral artery aneurysm (Vascular disorders) | 3 (4) | 3 (4)
Peripheral embolism (Vascular disorders) | 1 (1) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 3 (3)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endovascular Repair (N=444) | Open Repair (N=437)
Adynamic ileus (Gastrointestinal disorders) | 3 (3) | 22 (22) — AAA Related within 30 days
Agitation/anxiety (Psychiatric disorders) | 5 (5) | 19 (21) — AAA Related within 30 days
Anemia (Blood and lymphatic system disorders) | 7 (7) | 29 (29) — AAA Related within 30 days
Angina (Cardiac disorders) | 1 (1) | 0 (0) — AAA Related within 30 days
Arrhythmia (Cardiac disorders) | 3 (4) | 46 (51) — AAA Related within 30 days
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0) — AAA Related within 30 days
Bleeding complications (Injury, poisoning and procedural complications) | 3 (4) | 18 (19) — AAA Related within 30 days
Bowel ischemia (Gastrointestinal disorders) | 2 (3) | 5 (5) — AAA Related within 30 days
Branch vessel occlusion (Vascular disorders) | 0 (0) | 1 (1) — AAA Related within 30 days
Chest Pain (General disorders) | 0 (0) | 1 (1) — AAA Related within 30 days
Claudication (Vascular disorders) | 6 (10) | 1 (1) — AAA Related within 30 days
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 3 (4) — AAA Related within 30 days
Congestive Heart Failure (Cardiac disorders) | 2 (2) | 3 (3) — AAA Related within 30 days
Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 3 (4) — AAA Related within 30 days
Electrolyte imbalance (Metabolism and nutrition disorders) | 14 (16) | 55 (60) — AAA Related within 30 days
Embolism (Vascular disorders) | 1 (1) | 7 (7) — AAA Related within 30 days
Endoprosthesis migration or reallignment (General disorders) | 1 (2) | 0 (0) — AAA Related within 30 days
Endoprosthesis thrombosis (General disorders) | 2 (2) | 0 (0) — AAA Related within 30 days
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) — AAA Related within 30 days
Fever (General disorders) | 15 (16) | 16 (19) — AAA Related within 30 days
Hematoma (Vascular disorders) | 14 (14) | 4 (4) — AAA Related within 30 days
Hypertension (Vascular disorders) | 11 (13) | 20 (20) — AAA Related within 30 days
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — AAA Related within 30 days
Leg edema (General disorders) | 1 (1) | 10 (11) — AAA Related within 30 days
Lumen obstruction (Vascular disorders) | 2 (2) | 2 (2) — AAA Related within 30 days
Lymphocele (Vascular disorders) | 2 (2) | 2 (2) — AAA Related within 30 days
Myocardial Infarction (Cardiac disorders) | 2 (3) | 5 (5) — AAA Related within 30 days
Nerve injury (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) — AAA Related within 30 days
Pain (General disorders) | 61 (75) | 65 (75) — AAA Related within 30 days
Paraplegia/paraparesis (Nervous system disorders) | 1 (1) | 0 (0) — AAA Related within 30 days
Positive blood cultures (Investigations) | 0 (0) | 5 (5) — AAA Related within 30 days
Post operative nausea and vomiting (Injury, poisoning and procedural complications) | 13 (13) | 19 (19) — AAA Related within 30 days
Post-Implant syndrome (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — AAA Related within 30 days
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 4 (4) — AAA Related within 30 days
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — AAA Related within 30 days
Renal failure or other renal complications (Renal and urinary disorders) | 19 (23) | 36 (41) — AAA Related within 30 days
Respiratory complications (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 63 (83) — AAA Related within 30 days
Scrotal edema (Reproductive system and breast disorders) | 9 (9) | 3 (3) — AAA Related within 30 days
Troponin increase (Investigations) | 6 (6) | 17 (18) — AAA Related within 30 days
Vascular trauma (Injury, poisoning and procedural complications) | 0 (0) | 5 (5) — AAA Related within 30 days
Venous thrombosis (Vascular disorders) | 0 (0) | 3 (3) — AAA Related within 30 days
Wound infection (Infections and infestations) | 8 (8) | 11 (11) — AAA Related within 30 days
Other with no matching Adverse Event co (General disorders) | 38 (47) | 76 (125) — AAA Related within 30 days
Adynamic ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) — Not AAA Related within 30 days
Agitation/anxiety (Psychiatric disorders) | 0 (0) | 5 (5) — Not AAA Related within 30 days
Anemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) — Not AAA Related within 30 days
Arrhythmia (Cardiac disorders) | 4 (4) | 6 (6) — Not AAA Related within 30 days
Bowel ischemia (Gastrointestinal disorders) | 1 (1) | 0 (0) — Not AAA Related within 30 days
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) — Not AAA Related within 30 days
Chest Pain (General disorders) | 0 (0) | 1 (1) — Not AAA Related within 30 days
Coagulopathy (Blood and lymphatic system disorders) | 1 (2) | 1 (1) — Not AAA Related within 30 days
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 1 (1) — Not AAA Related within 30 days
Electrolyte imbalance (Metabolism and nutrition disorders) | 3 (3) | 5 (9) — Not AAA Related within 30 days
Fever (General disorders) | 8 (9) | 4 (4) — Not AAA Related within 30 days
Hematoma (Vascular disorders) | 1 (1) | 0 (0) — Not AAA Related within 30 days
Hypertension (Vascular disorders) | 0 (0) | 4 (4) — Not AAA Related within 30 days
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Not AAA Related within 30 days
Leg edema (General disorders) | 0 (0) | 1 (1) — Not AAA Related within 30 days
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) — Not AAA Related within 30 days
Pain (General disorders) | 6 (7) | 6 (7) — Not AAA Related within 30 days
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 3 (3) — Not AAA Related within 30 days
Renal failure or other renal complications (Renal and urinary disorders) | 5 (5) | 7 (7) — Not AAA Related within 30 days
Respiratory complications (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (13) — Not AAA Related within 30 days
Scrotal edema (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Not AAA Related within 30 days
Spinal neurological deficit (Nervous system disorders) | 0 (0) | 1 (1) — Not AAA Related within 30 days
Troponin increase (Investigations) | 1 (1) | 1 (1) — Not AAA Related within 30 days
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) — Not AAA Related within 30 days
Wound infection (Infections and infestations) | 1 (2) | 0 (0) — Not AAA Related within 30 days
Other with no matching Adverse Event co (General disorders) | 14 (21) | 24 (31) — Not AAA Related within 30 days
Access failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — AAA Related more than 30 days
Adynamic ileus (Gastrointestinal disorders) | 6 (6) | 9 (10) — AAA Related more than 30 days
Agitation/anxiety (Psychiatric disorders) | 3 (3) | 4 (4) — AAA Related more than 30 days
Amputation (Surgical and medical procedures) | 1 (1) | 2 (5) — AAA Related more than 30 days
Anemia (Blood and lymphatic system disorders) | 5 (5) | 6 (6) — AAA Related more than 30 days
Aneurysm enlargement (Vascular disorders) | 10 (15) | 1 (1) — AAA Related more than 30 days
Aneurysm rupture (Vascular disorders) | 2 (2) | 0 (0) — AAA Related more than 30 days
Arrhythmia (Cardiac disorders) | 7 (8) | 10 (11) — AAA Related more than 30 days
Bleeding complications (Injury, poisoning and procedural complications) | 4 (4) | 6 (7) — AAA Related more than 30 days
Bowel ischemia (Gastrointestinal disorders) | 2 (2) | 4 (5) — AAA Related more than 30 days
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 8 (9) — AAA Related more than 30 days
Branch vessel occlusion (Vascular disorders) | 2 (2) | 2 (3) — AAA Related more than 30 days
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (2) — AAA Related more than 30 days
Chest Pain (General disorders) | 0 (0) | 1 (1) — AAA Related more than 30 days
Chylous Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) — AAA Related more than 30 days
Claudication (Vascular disorders) | 8 (8) | 4 (4) — AAA Related more than 30 days
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) — AAA Related more than 30 days
Congestive Heart Failure (Cardiac disorders) | 0 (0) | 2 (2) — AAA Related more than 30 days
Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — AAA Related more than 30 days
Deployment failure (General disorders) | 1 (1) | 0 (0) — AAA Related more than 30 days
Electrolyte imbalance (Metabolism and nutrition disorders) | 7 (7) | 16 (19) — AAA Related more than 30 days
Embolism (Vascular disorders) | 2 (2) | 1 (1) — AAA Related more than 30 days
Endoprosthesis infection (Infections and infestations) | 4 (7) | 0 (0) — AAA Related more than 30 days
Endoprosthesis material failure or dilation (General disorders) | 2 (2) | 0 (0) — AAA Related more than 30 days
Endoprosthesis migration or reallignment (General disorders) | 11 (15) | 0 (0) — AAA Related more than 30 days
Endoprosthesis thrombosis (General disorders) | 8 (10) | 1 (1) — AAA Related more than 30 days
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 8 (9) — AAA Related more than 30 days
Fever (General disorders) | 5 (7) | 6 (6) — AAA Related more than 30 days
Hematoma (Vascular disorders) | 10 (11) | 1 (1) — AAA Related more than 30 days
Hypertension (Vascular disorders) | 5 (5) | 3 (4) — AAA Related more than 30 days
Incisional hernia (Injury, poisoning and procedural complications) | 5 (6) | 50 (69) — AAA Related more than 30 days
Leg edema (General disorders) | 5 (6) | 8 (8) — AAA Related more than 30 days
Lumen obstruction (Vascular disorders) | 7 (8) | 3 (3) — AAA Related more than 30 days
Lymphocele (Vascular disorders) | 5 (6) | 3 (3) — AAA Related more than 30 days
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) — AAA Related more than 30 days
Nerve injury (Injury, poisoning and procedural complications) | 5 (7) | 2 (2) — AAA Related more than 30 days
Pain (General disorders) | 20 (25) | 23 (31) — AAA Related more than 30 days
Paraplegia/paraparesis (Nervous system disorders) | 1 (1) | 0 (0) — AAA Related more than 30 days
Positive blood cultures (Investigations) | 0 (0) | 2 (5) — AAA Related more than 30 days
Post operative nausea and vomiting (General disorders) | 4 (4) | 4 (5) — AAA Related more than 30 days
Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — AAA Related more than 30 days
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 2 (7) — AAA Related more than 30 days
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — AAA Related more than 30 days
Renal failure or other renal complications (Renal and urinary disorders) | 20 (27) | 11 (15) — AAA Related more than 30 days
Respiratory complications (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 21 (29) — AAA Related more than 30 days
Scrotal edema (Reproductive system and breast disorders) | 2 (2) | 5 (6) — AAA Related more than 30 days
Troponin increase (Investigations) | 1 (1) | 5 (6) — AAA Related more than 30 days
Vascular trauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) — AAA Related more than 30 days
Venous thrombosis (Vascular disorders) | 1 (1) | 3 (3) — AAA Related more than 30 days
Wound infection (Infections and infestations) | 15 (18) | 13 (14) — AAA Related more than 30 days
Other with no matching Adverse Event co (General disorders) | 33 (43) | 44 (99) — AAA Related more than 30 days

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No